CLINICAL TRIAL: NCT00126113
Title: The Performance-Perceptual Test as a Counseling Tool
Acronym: PPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: C3951-R; 05-2504 (Other: Portland VA IRB); 11-2104 (Other: Portland VA IRB)
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Hearing Impairment
Keywords: Audiologic rehabilitation; Counseling
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPT-based Counseling (Experimental): Counseling based on Performance-Perceptual Discrepancy (PPDIS) consisting of explanation of hearing tests plus recommendations based on PPDIS
  Interventions: Behavioral: PPT-based Counseling
- Standard Educational Counseling (Other): Standard educational counseling consisting of explanation of hearing tests
  Interventions: Behavioral: Standard Educational Counseling

INTERVENTIONS:
Behavioral: PPT-based Counseling — Counseling based on Performance-Perceptual Discrepancy (PPDIS) consisting of explanation of hearing tests plus recommendations based on PPDIS
  Arms: PPT-based Counseling
Behavioral: Standard Educational Counseling — Standard educational counseling consisting of explanation of hearing tests
  Arms: Standard Educational Counseling

SUMMARY:
The purpose of the study is to determine whether a new test of ability to understand speech in noise and an associated counseling program can improve hearing aid satisfaction. Participants complete routine hearing tests, some hearing-related questionnaires and the new speech test. One group of participants receives the new form of counseling, the second group does not. Hearing aid satisfaction following 10 weeks hearing aid use is compared across the groups.

DETAILED DESCRIPTION:
Hearing aid dissatisfaction continues to be disappointingly high, even though hearing aid technology has improved dramatically over the last 10 years or so. Unfortunately, the results of most commonly used self-report measures cannot be directly compared with the results from performance measures since the modes of testing are very different. Thus, it is hard for clinicians to reconcile data from individuals reporting more handicap or less hearing aid satisfaction than would be expected from their performance.

In this study, the investigators use a test known as the Performance-Perceptual Test (PPT) to determine whether simple counseling based upon discussion of PPT results can be used to better align perceived and measured ability to understand speech-in-noise; and, more importantly, whether such counseling can decrease reported handicap and improve hearing aid satisfaction.

Hearing aid users complete the PPT for aided and unaided listening, along with standardized questionnaires measuring reported auditory disability, handicap and hearing aid satisfaction. Following this, subjects are randomly assigned to one of two groups. Subjects in Group 1 receive counseling from the experimenter in the form of an explanation and discussion of their PPT results. Subjects in Group 2 also participate in a discussion with the experimenter, but it does not include an explanation of the PPT. Two weeks after enrollment in the study subjects complete a second set of questionnaires. Ten weeks after study enrollment subjects return to the laboratory to rerun the test battery. The impact of the counseling upon PPT values, reported handicap and hearing aid satisfaction and benefit will be compared across the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate symmetrical sensorineural hearing loss
* Current users of binaural hearing aids

Exclusion Criteria:

* Conductive hearing impairment or other otological pathology
* A score less than age-based norms on the Mini Mental State Examination
* Asymmetrical hearing loss
* No prior use of hearing aids

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle H Saunders, Principal Investigator — VA Medical Center, Portland
Locations (1):
- VA Medical Center, Portland, Portland, Oregon, United States

REFERENCES:
- [Result] Saunders GH, Forsline A. Hearing-aid counseling: comparison of single-session informational counseling with single-session performance-perceptual counseling. Int J Audiol. 2012 Oct;51(10):754-64. doi: 10.3109/14992027.2012.699200. Epub 2012 Jul 19. PMID 22812927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dissatisfied hearing aid users recruited from Portland VA Medical Center Audiology Clinic. Recruitment dates: 1/1/06 to 9/1/07
Pre-assignment Details: Exclusion criteria were:
  Hearing aid dissatisfaction associated with physical fit of the hearing aids, conductive hearing loss, had not worn hearing aids for at least 3 months prior to participating, had mini mental status examination score below age and educationally-appropriate norms.
Period: Overall Study
Arm/Group | PPT-based Counseling | Standard Educational Counseling
Started | 37 | 37
Completed | 34 | 35
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PPT-based Counseling | Standard Educational Counseling | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.6) | 66.1 (7.8) | 65.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 34 | 32 | 66
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74
Hearing sensitivity (pure tone thresholds) [Mean (Standard Deviation); unit: decibels] | 45.0 (11.6) | 46.4 (11.0) | 45.7 (113)
Education level [Mean (Standard Deviation); unit: years] | 15.4 (3.1) | 15.1 (2.4) | 15.3 (2.8)
Past hearing aid use [Mean (Standard Deviation); unit: years] | 8.8 (10.3) | 9.8 (10.6) | 9.3 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Psychosocial Impact of Assistive Devices Scale (PIADS)
Description: PIADS: The PIADS measures the psychosocial impact of any assistive device(s). Here that is a hearing aid. The PIADS is a 26-item self-rating scale. The user rates each item on a seven-point scale that ranges from negative 3 (maximum negative impact) to positive 3 (maximum positive impact). The midpoint, zero, indicates no impact or no perceived change resulting from device use. It measures three quality-of-life domains: (1) Adaptability that reflects the inclination or motivation to participate socially and take risks; (2) Competence that reflects perceived functional capability, independence, and performance; and (3) Self-esteem that reflects self-confidence, self esteem, and emotional well-being.
Time Frame: Day 70 (end of study) only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PPT-based Counseling | Standard Educational Counseling
Number analyzed (Participants) | 34 | 35
units on a scale | 1.06 (0.79) | 0.85 (0.70)
Statistical Analysis 1: Comparison: PPT-based Counseling vs Standard Educational Counseling; Test type: Superiority or Other; p > 0.05, ANOVA; Analysis for main effect of group

2. Secondary Outcome: Hearing Handicap Inventory (HHI)
Description: HHI: The HHI for the elderly is for individuals over age 65 years; the HHI for adults is for individuals aged 65 years and younger. Both are 25-item questionnaires that assess the social and emotional consequences of hearing loss. The versions differ in the wording of three questions. Items are answered on a scale of Yes (4 points), Sometimes (2 points), and No (0 points) with higher scores indicating greater reported hearing handicap. Scores can range from 0 (no handicap) to 100 (maximum handicap).
Time Frame: Day 70 (end of study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PPT-based Counseling | Standard Educational Counseling
Number analyzed (Participants) | 34 | 35
units on a scale | 38.0 (19.4) | 34.7 (17.6)
Statistical Analysis 1: Comparison: PPT-based Counseling vs Standard Educational Counseling; Test type: Superiority or Other; p > 0.05, ANOVA — Analysis for main effect of group

3. Secondary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: APHAB: The APHAB is a 24-item questionnaire that documents hearing difficulties in specified listening situations. Items are answered on a seven-point scale from ' Always ' to ' Never ' with higher scores indicating greater reported hearing disability. The questionnaire has four subscales: Ease of communication, Reverberation, Background noise, and Aversiveness, from which a global score is computed by averaging the Ease of communication, Reverberation, and Background noise scale scores. Questions are answered for unaided and aided listening. By subtracting aided scores from unaided scores a measure of reported aided benefit is obtained. Scores can range from 0 (no disability) to 99 (maximum disability).
Time Frame: Day 70 (end of study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PPT-based Counseling | Standard Educational Counseling
Number analyzed (Participants) | 34 | 35
units on a scale | 26.3 (15.2) | 21.9 (14.8)
Statistical Analysis 1: Comparison: PPT-based Counseling vs Standard Educational Counseling; Test type: Superiority or Other; p > 0.05, ANOVA; Analysis for main effect of group

4. Secondary Outcome: International Outcome Inventory for Hearing Aids (IOI-HA)
Description: The IOI-HA is a seven-item questionnaire for which hearing-aid use, hearing-aid benefit, residual activity limitation, hearing-aid satisfaction, residual participation restriction, impact on others, and quality of life are rated on a five-point scale. An overall IOI-HA score is generated by averaging responses to all seven items. Higher scores reflect better self-reported outcome. Scores can range from 7 (poorest outcome) to 35 (best outcome).
Time Frame: Day 70 (end of study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PPT-based Counseling | Standard Educational Counseling
Number analyzed (Participants) | 34 | 35
units on a scale | 26.6 (4.2) | 25.5 (4.8)
Statistical Analysis 1: Comparison: PPT-based Counseling vs Standard Educational Counseling; Test type: Superiority or Other; p > 0.05, ANOVA; Analysis for main effect of group

ADVERSE EVENTS:
Arm/Group | PPT-based Counseling | Standard Educational Counseling
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No